CLINICAL TRIAL: NCT06671431
Title: Role of Adjuvant Chemotherapy in Distal Cholangiocarcinoma: a Retrospective Cohort Study
Brief Title: Role of Adjuvant Chemotherapy in Distal Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2408-168-1565
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Distal Cholangiocarcinoma; Adjuvant Chemotherapy
MeSH Terms: interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Adjuvant chemotherapy — Adjuvant chemotherapy with or without radiotherapy

SUMMARY:
Recent studies addressing the role of adjuvant chemotherapy in cholangiocarcinoma (CCA) have been published; however, there are challenges in generalizing the findings due to different prognostic characteristics depending on tumor location and resectability. Therefore, the aim of this study was to investigate the role of AC in distal cholangiocarcinoma, a common tumor subtype of CCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal cholangiocarcinoma who underwent surgery

Exclusion Criteria:

* Who underwent neoadjuvant treatment
* Who underwent R2 resection
* Non-adenocarcinoma patients in final pathology report
* Insufficient data
* Death within 90days of surgery

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with distal cholangiocarcinoma who underwent curative surgery
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Role of Adjuvant Chemotherapy in Distal Cholangiocarcinoma | From January 2000 to December 2021